CLINICAL TRIAL: NCT01384695
Title: A Feasibility Study of Confocal Microendoscopy in the Evaluation of Gastrointestinal Neoplasia - Project 1
Brief Title: A Feasibility Study of Confocal Microendoscopy in the Evaluation of Gastrointestinal Neoplasia -Project 1
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Low/no enrollment. No subjects were enrolled over the past year.
Sponsor: Anandasabapathy, Sharmila, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: GCO# 09-0696 Project 1
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: GERD; Barrett's Esophagus
Keywords: Barrett's esophagus; confocal microendoscopy
MeSH Terms: conditions — Gastroesophageal Reflux; Barrett Esophagus | interventions — Fluorescein; Proflavine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluorescein (Experimental): Confocal imaging using contrast agent fluorescein
  Interventions: Drug: Proflavine hemisulfate
- Proflavine hemisulfate (Experimental): confocal imaging using contrast agent proflavine
  Interventions: Drug: Fluorescein

INTERVENTIONS:
Drug: Fluorescein — fluorescent contrast agent, Fluorescein 5ml
  Arms: Proflavine hemisulfate
Drug: Proflavine hemisulfate — 3 ml of 0.01% proflavine (derived from dissolving 10mg proflavine hemisulfate USP in 100ml sterile water)
  Other Names: Proflavine
  Arms: Fluorescein

SUMMARY:
The overall objective of this study is to obtain data to evaluate whether high-resolution imaging of the gastrointestinal mucosain vivo can assist clinicians in detecting dysplastic (precancerous) areas. This is an exploratory study of a confocal endoscope designed to evaluate the feasibility of using this FDA-approved device in the endoscopic surveillance of subjects at high-risk for neoplasia in the upper and lower GI tract. The confocal endoscope provides real-time in vivo microscopic images of the mucosa which resemble standard pathology.

ELIGIBILITY:
Inclusion Criteria:

* patient 18 years or older
* colonoscopy for screening or surveillance of polyps or disease of colon
* anoscopy because of suspected or known anal dysplasia or neoplasia

Exclusion Criteria:

* patient unable to provide informed consent
* patient found unfit for standard colonoscopy or anoscopy with biopsies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2009-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
to determine whether tissue is neoplastic or non-neoplastic | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Anandasabapathy, M.D., Principal Investigator — Mt. Sinai School of Medicine
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States